CLINICAL TRIAL: NCT04298489
Title: Personalized Drug Sensitivity Test for Late Stage, Potentially Operable Gastrointestinal Cancer Using Patient Derived Primary Cell Culture
Brief Title: Drug Sensitivity Screening for Gastrointestinal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Aiwen Wu, M.D. PH.D. Chief, Unit III & Ostomy Service, Gastrointestinal Cancer Center, Peking University Cancer Hospital & Institute, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PKUCH-M01
Record Dates: First submitted 2018-12-10; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Gastrointestinal Cancer Metastatic
Keywords: Personalized; Drug Sensitivity Test; Chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stage III/IV gastrointestinal cancer patients (Experimental): The study group (Personalized drug sensitivity test) was treated according to the physician's opinion. Tumor tissues are obtained during the surgery or via biopsy with informed consent, for the purpose of ex vivo assay.
  Interventions: Diagnostic Test: Personalized drug sensitivity test

INTERVENTIONS:
Diagnostic Test: Personalized drug sensitivity test — The patients underwent surgery to remove tumor and took out tumor specimens for research. The tumor cells were expanded ex vivo drug sensitivity assay.
  The drugs used in the study were 5-fluorouracil, Oxaliplatin, and irinotecan at C0 = 10 mM, 2.5 mM and 0.02 mM, respectively. They were applied either as single agents or in combinations of 5-fluorouracil and Oxaliplatin, 5-fluorouracil and irinotecan, or all three agents, or others. After 7 days of treatment, the tumor cells were stained with EdU, Hoechst and EpCAM with the Cell Quantitative Detection Kit. Images were acquired with an automated microscopic image-scanning system and analyzed with the built-in software.

SUMMARY:
Explore the clinical feasibility of using primary cell culture system to guide gastrointestinal cancer chemotherapy, and establish the correlation between ex vivo drug sensitivity and patient clinical response.

Study objectives: Personalized drug sensitivity test for late stage,potentially operable gastrointestinal cancer using patient derived primary cell culture.

Explore the clinical feasibility of using primary cell culture system to guide gastrointestinal cancer chemotherapy, and establish the correlation between ex vivo drug sensitivity and patient clinical response.

The study will collect primary tumor tissues from stage III/IV gastrointestinal cancer patients who underwent emergency surgeries, and then establish the primary tumor cell library for ex vivo chemotherapy drug sensitivity test in order to:

1. Compare the ex vivo Maximal Inhibition Index(MI) and Drug Sensitivity Index (DSI) with patient's Overall Response Rate (ORR)
2. Provide research support for future clinical treatment.

This ex vivo method applies to single or combination drug regimen, and does not require prior knowledge of the specific mechanism for individual patient's drug sensitivity. Previous research as well as literature studies support the close relationship between ex vivo drug sensitivity and in vivo drug response.

DETAILED DESCRIPTION:
The patient underwent surgery to remove tumor and agreed to take out the abdominal tumor specimens for research. A section of each sample was removed for the generation of PDX models as described early.The rest of the tumor cells were expanded using ex vivo drug sensitivity assay.

The drugs used in the study were 5-fluorouracil, Oxaliplatin, and irinotecan at C0 = 10 mM, 2.5 mM and 0.02 mM, respectively. They were applied either as single agents or in combinations of 5-fluorouracil and Oxaliplatin, 5-fluorouracil and irinotecan, or all three agents, or others. After 7 days of treatment, the tumor cells were stained with EdU, Hoechst and EpCAM with the Cell Quantitative Detection Kit. Images were acquired with an automated microscopic image-scanning system and analyzed with the built-in software.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients between 18 and 70 years old, male or female;
2. Voluntary patient consent；
3. Treatment-naïve, stage III/IV gastrointestinal cancer patients with pathology confirmation；
4. According clinical researcher, patient has operable tumor lesion, and tumor tissue can be obtained through surgical removal;
5. Good tolerability to standard chemotherapy regimen；
6. ECOG status <3；
7. Estimated survival time no less than 6 months；
8. Patient has at least one measurable disease lesion (according to RECIST1.1).

Exclusion Criteria:

1. Patient has received any prior anti-cancer treatment;
2. Participated in any other clinical study within 6 months;
3. Women currently breast feeding or pregnant;
4. Severe liver or kidney function impairment (Live function: TBIL ≤1.5×ULN，ALT & AST≤2.5×ULN);
5. Patients with liver metastasis ≤5.0×ULN；Kidney function：Cr ≤1.5×ULN and creatinine clearance rate≥ 50 mL/min (according to the Cockcroft-Gault formula);
6. Patients with cognitive impairment, psychological disease, or poor compliance;
7. Allergic to known chemotherapy ingredients;
8. Other factors researchers deemed not suitable for study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
ex vivo Maximal Inhibition Index (MI) | 1 month after the tissue acquisition
  The effectiveness of each therapeutic regimen was evaluated and quantified using the formula: Maximum Inhibition (MI)=N0/Nd, where N0 and Nd denotes the number of EpCAM+ EdU+ epithelial cells in the wells of control or withthe drug at concentration C0, respectively.

SECONDARY OUTCOMES:
Disease Control Rate（DCR）after chemotherapy | 3 months after chemotherapy
  Disease Control Rate（DCR）after chemotherapy.
Progression free survival (PFS) after chemotherapy | 1 year after chemotherapy
  Progression free survival (PFS) after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Aiwen Wu, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China